CLINICAL TRIAL: NCT06851923
Title: Study of Visual Mecanisms Involved in Face Recognition
Acronym: HUMVIS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HUMVIS
Record Dates: First submitted 2025-02-07; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Young Healthy Adults; Healthy
Keywords: face perception; Magnetic Resonance Imaging; 3 Tesla; human vision; orientation selectivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study of the visual mechanisms involved in face perception (Experimental)
  Interventions: Other: 3Tesla magnetic resonance imaging of the healthy human visual system

INTERVENTIONS:
Other: 3Tesla magnetic resonance imaging of the healthy human visual system — The present project presents a series of monocentric MRI studies carried out on healthy adult human volunteers. All neuroimaging will be performed at the Cliniques Universitaires Saint-Luc (CUSL, IRM de recherche). Participants will not directly benefit from their participation. All studies will manipulate the visual properties of the experimental stimuli in a within-subject way, and therefore do not rely on any participation group assignation/randomization method. The duration of studies will vary between 3h to 6h, i.e., from 2 to 4x1h30 3Tesla magnetic resonance imaging sessions depending on the experimental design.

SUMMARY:
Since the 19th century, perception has been regarded as an inferential process in which sensory input is compared with prior knowledge, namely the internalised representation of the visual environment. This notion is central to the understanding of everyday perception and cognition in general, and is attracting much attention in various areas of psychology and cognitive neuroscience. However, it is unclear whether and how the primary visual refinement that is thought to underlie the convergence of bottom-up inputs with top-down prior knowledge applies to the processing of meaningful stimuli in our everyday lives. The investigators have shown that human face processing mechanisms are shaped by prior knowledge that the horizontal range of face information conveys the richest and most reliable cues. Furthermore, investigators' previous data suggest that the primary visual cortex is recruited during the progressive refinement of face representation. Using very high field neuroimaging, the present project proposes to follow the neural mechanisms underlying the cortical refinement of horizontal information in human face processing, and to study their contribution to behaviour.

ELIGIBILITY:
Inclusion Criteria:

Participants will be screened (see annex 2) to ascertain they fit with all these inclusion criteria:

* Be between 18 and 50 years old,
* have normal eyesight or eyesight corrected with contact lenses,
* Have no neurological disorder,
* Not have had a skull fracture or head surgery,
* Have no chronic progressive illness or mental deficiency,
* Have no metal parts in their body (dental braces or pins, metal plates, pacemakers, implanted prostheses, etc.),
* Have no tattoos containing metallic particles or implanted jewellery (e.g. piercings) that cannot be removed,
* Not to have worked with metals,
* Do not take any medicines or substances that may affect brain function (e.g. drugs, energy drinks, alcohol),
* Not to be pregnant or breastfeeding.
* Do not be claustrophobic.

Exclusion Criteria:

Participants presenting a counter-indication (responding yes to one of the questions of the screening questionnaire, see annex 2) to participate will be excluded from participation.

Participants will be screened to ascertain they do not present any of these counter-indications to the participation to the MRI measurement. We will exclude people with these characteristics:

* Be younger than 18 or older than 50 years old,
* have poor eyesight,
* Have neurological disorder,
* have had a skull fracture or head surgery,
* Have a chronic progressive illness or mental deficiency,
* Have metal parts in their body (dental braces or pins, metal plates, pacemakers, implanted prostheses, etc.),
* Have tattoos containing metallic particles or implanted jewellery (e.g. piercings) that cannot be removed,
* have worked with metals,
* take medicines or substances that may affect brain function (e.g. drugs, energy drinks, alcohol),
* pregnant or breastfeeding.
* claustrophobic.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2030-11-15 (Estimated); Study Completion 2030-11-15 (Estimated)

PRIMARY OUTCOMES:
Orientation tuning in the visual system | 2 years
  fMRI will be used to analyse brain responses along the ventral visual pathway to the visual presentation of orientation-filtered visual face and scene stimuli
Emergence of orientation tuning over processing course in the visual system | 2 years
  fMRI will be used to analyse brain responses along the ventral visual pathway to the visual presentation of temporally masked orientation-filtered visual stimuli
Receptive field mapping of the visual system | 2 years
  fMRI will be used to measure population receptive fields using stimuli varying in position and size randomly
Behavioral task performance | 2 years
  Participants will identify famous faces presented on-screen and respond via keypress.

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Goffaux, PhD, Study Director — Université Catholique de Louvain; Mrittika Dey, Master, Principal Investigator — Université Catholique de Louvain

IPD SHARING:
Plan to Share IPD: No